CLINICAL TRIAL: NCT00416780
Title: Psychobiological Pathways: Breast Cancer Interventions
Brief Title: Psychosocial Support in Treating Women With Recurrent Breast Cancer or Stage I, Stage II, or Stage IV Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pittsburgh Mind-Body Center at Carnegie Mellon University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: PMBC-HS05-182; CMU-00000603 (Other: cmu); MWH-99-062; CDR0000459773 (Registry Identifier: PDQ (Physician Data Query)); FWA00004206
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2006-03

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

INTERVENTIONS:
Other: counseling intervention
Other: educational intervention
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Meeting together with other breast cancer patients to receive psychosocial support and to learn to reduce stress may help patients cope with their diagnosis, have a better quality of life, and live more comfortably.

PURPOSE: This randomized clinical trial is studying how well psychosocial support works in treating women with recurrent breast cancer or stage I, stage II, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate theoretically derived psychosocial interventions (peer discussion support vs education and stress management vs usual-care control) targeted to enhance adjustment and functional status and lower morbidity among women diagnosed with and treated for recurrent or stage I, II, or IV breast cancer.
* Evaluate the psychological, behavioral, and biological pathways and their effects in patients treated with these interventions.
* Evaluate the efficacy of these intervention in these patients.
* Evaluate the nature and extent of coping strategies in these patients.
* Evaluate the differences in patients treated with these intervention vs those patients electing not to be treated with these interventions.

OUTLINE: This is a randomized study. Patients are stratified according to disease stage (early vs late). Patients with early-stage disease are randomized to 1 of 3 intervention arms. Patients with late-stage disease are randomized to 1 of 2 intervention arms (II or III).

* Arm I (education and stress management): Patients undergo a 1-hour group (6-10 patients per group) education session once a week for 8 weeks focusing on exchange of factual information between a facilitator and patients. The session includes a 45-minute lecture, discussing risks, diagnosis, and treatment of cancer; side effects from treatment; nutrition during treatment; and follow-up care, followed by a question/answer period and instruction in progressive relaxation techniques. Patients then receive 3 monthly phone calls from a project staff member to answer questions about cancer, treatment, and follow-up care and to discuss the relaxation exercises.
* Arm II (peer discussion): Patients undergo a 1-hour group (6-10 patients per group) peer support session once a week for 8 weeks focusing on the provision of emotional support among patients and the maintenance of purpose in life. The session emphasizes on the sharing of experiences, the development of a common bond, and the promotion of altruism to similar others. Patients then are given an opportunity to attend 3 monthly additional meetings to share critical experiences and problems they have experienced in the past month.
* Arm III (control): Patients receive usual care and are not asked to attend any meetings.

All patients undergo a 2-hour baseline interview, a 1.5-hour post intervention interview, and a 1.5-hour final interview 8 months after randomization.

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with breast cancer

  * First-time diagnosis of stage I or II disease

    * No more than 2 months since prior breast cancer surgery
  * Initial diagnosis of stage IV disease
  * Distant recurrence of prior breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Reside within a 60-mile radius of the greater Pittsburgh metropolitan area

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scheier, PhD, Study Chair — Pittsburgh Mind-Body Center at Carnegie Mellon University